CLINICAL TRIAL: NCT03653416
Title: Comparison Between Ipack Block and Periarticular Infiltration in Total Knee Arthroplasty - a Randomized Control Trial
Brief Title: Efficacy of Ipack Block and Surgeon's Joint Infiltration in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Yan Lai, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 17-04304; IRB 17-01981 (Other: PPHS, ISMMS)
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Results first posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Osteo Arthritis Knee
Keywords: Total knee arthroplasty; Peri articular infiltration; Pack block; Adductor canal catheter
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Ipack group (Experimental): 20 cc of bupivacaine(o.25%) will be injected with the help of ultrasound guidance. Patients will receive adductor canal catheter and peri articular infiltration as well.
  Interventions: Device: Ipack; Drug: Bupivacaine; Procedure: Peri Articular Infiltration
- Pai (peri articular) group (Active Comparator): Patients will receive adductor canal catheter and peri articular infiltration.
  Interventions: Procedure: Peri Articular Infiltration

INTERVENTIONS:
Device: Ipack — IPACK block - local anesthesia injected safely under ultrasound guidance in the interspace between the popliteal artery and capsule of the knee.
  Arms: Ipack group
Drug: Bupivacaine — 20 cc of bupivacaine(o.25%) injection
  Arms: Ipack group
Procedure: Peri Articular Infiltration — Adductor Canal Catheter and Peri Articular Infiltration
  Other Names: PAI

SUMMARY:
Total knee arthroplasty(TKA) is an effective modality for the treatment of advanced osteoarthritis of the knee joint with excellent outcomes. With 719,000 cases being performed as of 2010, the incidence is expected to increase up to 3.48 million procedures annually by 2030.

DETAILED DESCRIPTION:
There have been several studies regarding efficacy of peri articular infiltration. IPACK block is a novel technique gaining popularity where one injects local anesthesia safely under ultrasound guidance in the interspace between the popliteal artery and capsule of the knee.

There have been no studies till date comparing the efficacy between IPACK block and Periarticular Infiltration (PAI).

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiology) class I-IV
* age 18-75.

Exclusion Criteria:

* ASA class V
* morbid obesity
* patient refusal
* patients with chronic pain or on pain medication
* allergy to LA
* patients receiving any additional regional techniques
* coagulopathy
* patients receiving systemic anticoagulation
* local infection and procedures anticipated to last more than 5 hours.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 99 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan H Lai, MD,MPH, Principal Investigator — Ichan School of Medicine
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sankineani SR, Reddy ARC, Eachempati KK, Jangale A, Gurava Reddy AV. Comparison of adductor canal block and IPACK block (interspace between the popliteal artery and the capsule of the posterior knee) with adductor canal block alone after total knee arthroplasty: a prospective control trial on pain and knee function in immediate postoperative period. Eur J Orthop Surg Traumatol. 2018 Oct;28(7):1391-1395. doi: 10.1007/s00590-018-2218-7. Epub 2018 May 2. PMID 29721648
- [Derived] Bh PP, Jinadu S, Okunlola O, Darkzali H, Lin HM, Lai YH. Integrating IPACK (Interspace between the Popliteal Artery and Capsule of the Posterior Knee) Block in an Enhanced Recovery after Surgery Pathway for Total Knee Arthroplasty-A Prospective Triple-Blinded Randomized Controlled Trial. J Knee Surg. 2023 Oct;36(12):1289-1296. doi: 10.1055/s-0042-1755355. Epub 2022 Aug 9. PMID 35944566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from March 2018, and study conducted from June 2018 to August 2019
Groups:
- Ipack Group: 20 cc of bupivacaine(o.25%) injected with the help of ultrasound guidance. Patients received adductor canal catheter and peri articular infiltration as well.
  Ipack: IPACK block - local anesthesia injected safely under ultrasound guidance in the interspace between the popliteal artery and capsule of the knee.
- Pai (Peri Articular) Group: Patients received adductor canal catheter and peri articular infiltration.
Period: Overall Study
Arm/Group | Ipack Group | Pai (Peri Articular) Group
Started | 52 | 47
Completed | 46 | 46
Not Completed | 6 | 1
Not completed — Protocol Violation | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pai (Peri Articular) Group | Ipack Group | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.65 (6.20) | 64.67 (7.72) | 63.66 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 14 | 44
  Male | 16 | 32 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 20 | 10 | 30
  Black or African American | 10 | 20 | 30
  Hispanic or Latino | 10 | 6 | 16
  White | 6 | 10 | 16
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.69 (7.27) | 31.74 (6.34) | 32.21 (6.80)
Side of surgery [Count of Participants; unit: Participants]
  Left | 20 | 20 | 40
  Right | 26 | 26 | 52
Smoker [Count of Participants; unit: Participants] | 1 | 5 | 6
Alcohol Use [Count of Participants; unit: Participants] | 16 | 13 | 29
Education Level [Count of Participants; unit: Participants]
  High School | 24 | 29 | 53
  Bachelor's degree | 12 | 11 | 23
  Graduate degree | 10 | 6 | 16
Number of Employed Participants [Count of Participants; unit: Participants] | 16 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Narcotic Consumption
Description: Narcotic consumption in the first 24 hours
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: morphine equivalents, mg
Arm/Group | Ipack Group | Pai (Peri Articular) Group
Number analyzed (Participants) | 46 | 46
morphine equivalents, mg | 15.87 (19.75) | 13.67 (19.39)

2. Secondary Outcome: Visual Analogue Score (VAS) for Pain
Description: Visual Analogue Score (VAS) for pain - scored from 0 (no pain) to 10 (extreme pain), that is, higher score indicates more pain.
Time Frame: at 6, 12, 18, and 24 hours post procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ipack Group | Pai (Peri Articular) Group
Number analyzed (Participants) | 46 | 46
score on a scale
  6 hours | 0.93 (2.05) | 0.93 (2.19)
  12 hours | 0.76 (1.62) | 0.93 (2.19)
  18 hours | 0.74 (1.93) | 1.41 (2.21)
  24 hours | 1.50 (2.53) | 2.18 (2.51)

3. Secondary Outcome: Time to First Dose of Narcotic Administration
Time Frame: up to 24 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Ipack Group | Pai (Peri Articular) Group
Number analyzed (Participants) | 46 | 46
hours | 1.5 [0.00 to 7.00] | 0.25 [0.00 to 4.00]

4. Secondary Outcome: PACU Length of Stay
Description: Post-Anesthesia Care Unit (PACU) length of stay (LOS)
Time Frame: average 24 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Ipack Group | Pai (Peri Articular) Group
Number analyzed (Participants) | 46 | 46
hours | 3.00 [2.50 to 4.51] | 3.00 [3.00 to 5.00]

5. Secondary Outcome: Number of Participants With Pain by Location
Description: Location of knee pain as anterior/posterior, medial/lateral
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ipack Group | Pai (Peri Articular) Group
Number analyzed (Participants) | 46 | 46
Participants
  Anterior | 1 | 0
  Knee | 4 | 18
  Lateral | 10 | 7
  Medial | 5 | 3
  Posterior | 4 | 18
  No Pain | 22 | 0

6. Secondary Outcome: Ambulation Distance
Description: Ambulation distance with assistance on Post-operative Day (POD) 1 as assessed by PT
Time Frame: Post-op Day 1
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Ipack Group | Pai (Peri Articular) Group
Number analyzed (Participants) | 46 | 46
meters | 50 [30 to 74] | 45 [15 to 100]

7. Secondary Outcome: Bartels Index
Description: Bartels Index to measure activities of daily living (ADL's) on POD 1 as assessed by OT. Total possible scores range from 0-100, with higher scores indicating more independence.
Time Frame: Post-op Day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ipack Group | Pai (Peri Articular) Group
Number analyzed (Participants) | 46 | 46
score on a scale | 47 [38 to 53] | 39 [38 to 53]

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Ipack Group | Pai (Peri Articular) Group
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT03653416/Prot_SAP_000.pdf